CLINICAL TRIAL: NCT06098768
Title: Effectiveness of Parent Led Implementation of a Virtual Reality Social Skills Training Program for Children With Autism Spectrum Disorder
Brief Title: Parent Led Implementation of a VR Social Skills Training Program for Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West Virginia University (Other)
Collaborators: Floreo (Unknown)
Responsible Party: Principal Investigator, Krestin Radonovich, Vice Chair of Research, Director of Pediatric Neuropsychology, West Virginia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2304763205
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Floreo BSC (Other): Subjects and their caregiver will engage in the Floreo VR Building Social Connections VR sessions: three sessions per week, for 12 weeks. Each session will consist of 2 VR (Floreo BSC) lessons separated by a brief break, for a total of approximately 15 minutes of direct VR time over a 30-minute period. Treatment sessions will be scheduled over a 12-week period, with an allowance of up to 15 weeks for make-up sessions (e.g., illness or travel).
  Interventions: Behavioral: VR Social Skills

INTERVENTIONS:
Behavioral: VR Social Skills — The intervention will consist of two episodes of the Floreo BSC program, each lasting 4-5 minutes, according to a fixed program of episodes determined by the participant's color-coded group. VR episodes will be presented via the Floreo application downloaded onto an iPhone worn by the participant in the VR headset. The VR interaction will be controlled and operated via linked iPad.

SUMMARY:
The goal of this interventional trial is to establish training protocols to show feasibility of training parents and caregivers to administer the VR protocol. The primary objective is to evaluate the effects of treatment with Floreo Building Social Connections (BSC) on the AIM, a parent report survey that assesses core symptoms of ASD. The secondary objective is to explore the changes in social skills over time by using a multimethod outcomes battery. The Investigators will evaluate the effect of treatment with Floreo BSC on the Childhood Autism Rating Scales (CARS-2) in the study patient population. Additional secondary objectives include evaluation of the effects of treatment on adaptive skills as measured by the Vineland-3. Participants will be asked to complete questionnaires and utilize the VR program at clinic and at home.

ELIGIBILITY:
Inclusion Criteria:

* Patients or legally authorized representatives must provide written informed consent and be willing and able to comply with study procedures. Participants must provide informed assent as clinically appropriate.
* A diagnosis of autism spectrum disorder on the basis of the clinical judgement of a qualified clinician according to DSM-5 criteria, supported by either the Autism Diagnostic Observation Schedule or the Autism Diagnostic Interview-Revised.
* Participants must be able to tolerate VR therapy in the judgement of parent or caregiver and study staff.
* Female participants must either be unable to become pregnant (e.g., premenarchal, surgically sterile, etc.) or agree to use a highly effective method of contraception (e.g., intrauterine device, oral contraceptives, condom or diaphragm with spermicides, contraceptive sponge) from 28 days before the Baseline Visit to 45 days after the last treatment session. Females of childbearing potential must have a negative urine human chorionic gonadotropin pregnancy test at the Screening Visit.

Exclusion Criteria:

* History of photosensitive epilepsy or demonstrated photoparoxysmal response on prior electroencephalogram.
* Active diagnosis of migraine headache or migraine variant (abdominal migraine, cyclic vomiting syndrome) which is not adequately controlled by medication or other therapy.
* History of balance disorder including vertigo, motion sensitivity, or ataxia. Vestibular sensory deficits are not necessarily exclusionary.
* Primary sensory impairment (blindness, deafness).
* Motor disorder that would interfere with VR engagement.

Ages: 4 Years to 131 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Autism Impact Measure (AIM) | Baseline to 1 week post final treatment visit
  Change in measure: The AIM is a 25-item parent questionnaire targeting sensitivity to change of core ASD symptoms (Kanne et al., 2014). The questionnaire uses a 2-week recall period with items rated on two corresponding 5-point scales (frequency and impact). 5-point Likert-type scale, once for frequency of a specific behavior of the dependent and once for impact of that behavior. Response options range from "never" to "always" for the frequency dimension and "not at all" to "severely" for the impact dimension. Higher domain and higher total scores indicate greater symptom severity (Houghton et al., 2019; Mazurek et al., 2018). Likewise, lower AIM scores indicate less severe symptomatology.
Childhood Autism Rating Scale, 2nd Edition (CARS-2) | Baseline to 1 week post final treatment visit
  Change in score from Baseline up to 1 week post final treatment visit. The CARS2 total raw score range from 15 to 60. This scale is a behavior rating scale intended to diagnose autism. A total score of 15 indicates that an individual behavior is within normal limits, whereas a value of 60 indicates that the individual's behavior is severely abnormal.
Vineland Scales of Adaptive Behavior, 3rd Edition (Vineland 3) | Baseline to 1 week post final treatment visit
  Change in Measure for The Vineland-3 which evaluates adaptive behavior in five different domains: Social, Communication, Daily Living Skills, and Motor (Sparrow et al., 2016). In the context of this study, it will be administered using the Comprehensive Interview Form, for which a parent or caregiver is interviewed by a qualified rater familiar with the instrument. Based on the summarized scores in each domain, an Adaptive Behavior Composite (ABC) is also calculated. Items are scored on a scale of 0 (never), 1 (sometimes), or 2 (usually) for the level at which the child can independently perform a skill. The higher the score, the better the adaptive level.

CONTACTS AND LOCATIONS:
Overall Officials: Krestin Radonovich, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States